CLINICAL TRIAL: NCT01267799
Title: Correlation Between Pulmonary Function and Selected Serum/Sputum Biomarkers of Pulmonary Damage Among Workers in Photocopier Units
Brief Title: Health Status of Workers in Photocopier Units
Status: Completed | Type: Observational
Sponsor: Avinashilingam Deemed University (Other)
Responsible Party: Principal Investigator, E. Nithya, Research Scholar, Avinashilingam Deemed University
Other Study IDs: photocopiers
Record Dates: First submitted 2010-12-28; First posted 2010-12-29 (Estimated); Last update posted 2017-06-29 (Actual); Status verified 2017-06

CONDITIONS: Exposure to Photocopiers on a Professional Basis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- photocopier exposure
- control

SUMMARY:
Photocopiers are indispensable in today's working environment. However, photocopiers emit a number of harmful chemicals during their operation. Photocopier toners also contain a number of potentially toxic substances. Chronic exposure to these substances may compromise the health of photocopier operators. This study is aimed to understand if chronic exposure to photocopier emissions is harmful to human health.

ELIGIBILITY:
Inclusion Criteria:

Exposure to photocopier emissions for minimum 2 years professionally

Exclusion Criteria:

Any clinical abnormality

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: exposure to photocopier emissions
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2011-07 (Actual); Primary Completion 2012-07 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
To assess if photocopier emissions are toxic to human health | 2 years

SECONDARY OUTCOMES:
To assess the best biomarker for pulmonary damage in serum | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jeyanthi G P, Ph.D, Study Director — Avinashilingam Deemed University for Women
Locations (3):
- India (3):
  - Avinashilingam Deemed University for Women, Coimbatore, Tamil Nadu
  - Avinashilingam Deemed University, Coimbatore, Tamil Nadu
  - Coimbatore, Tamil Nadu